CLINICAL TRIAL: NCT01899066
Title: Lucentis in the Treatment of Retinoblastoma - A Phase II, Single Center, Randomized Study to Evaluate the Efficacy of Ranibizumab in Subjects With Retinoblastoma
Brief Title: Efficacy Study of Lucentis in the Treatment of Retinoblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Efficacy Study of Lucentis in the Treatment of Retinoblastoma, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yanghs20130627
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Retinoblastoma
Keywords: Efficacy
MeSH Terms: conditions — Retinoblastoma | interventions — Ranibizumab; Drug Therapy; Vincristine; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lucentis; chemotherapy (Experimental): Lucentis: 0.5mg/0.05 ml;Other Name: Ranibizumab;monthly for the first six months.
  Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months.
  Interventions: Drug: Lucentis, chemotherapy
- chemotherapy (Active Comparator): chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: Lucentis, chemotherapy — Lucentis:0.50mg/0.05ml, intravitreal injection,monthly for the first six months.
  chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.
  Other Names: Ranibizumab
  Arms: Lucentis; chemotherapy
Drug: chemotherapy — chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.
  Other Names: vincristine;; carboplatin;; etoposide.
  Arms: chemotherapy

SUMMARY:
This study will evaluate the clinical efficacy of intravitreal injections of Ranibizumab (Lucentis) together with chemotherapy in the treatment of Retinoblastoma as compared to chemotherapy alone.

DETAILED DESCRIPTION:
This study will be a phase II open label interventional case series. Patients with retinoblastoma will be randomized to receive chemotherapy with or without intravitreal ranibizumab at a dose of 0.5mg/0.05 ml. Patients will receive ranibizumab via a pars plana injection on a monthly basis for a total duration of therapy of 6 months. Patients will be followed for 24 months .

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Definite characteristic signs of retinoblastoma,Group D base on Intraocular International Retinoblastoma classify, IIRC.

Exclusion Criteria:

* History of surgical intervention for retinoblastoma in the study eye.
* Any previous disease in the study eye.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).
* Previous participation in a clinical trial (for either eye) involving anti angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two years
  measure the mortality rate for the two groups(Cancer-related death and non-Cancer-related death) at two years

SECONDARY OUTCOMES:
Efficacy of Lucentis(intravitreal injection) in the Treatment of Retinoblastoma | two years
  measure the tumor size and new vessels by ultrasonography，fundus photography and fundoscopy before each treatment, and 1,3,6,9,12,18,24 months after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, Study Chair — Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China